CLINICAL TRIAL: NCT00878826
Title: Prophylactic Enoxaparin Dosing for Prevention of Venous Thromboembolism in Pregnancy.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Deirdre Judith Lyell, Associate Professor, Obstetrics and Gynecology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SU-03172009-2003; 15957 (Other: Stanford University IRB)
Record Dates: First submitted 2009-04-07; First posted 2009-04-09 (Estimated); Results first posted 2013-09-05 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-10

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Enoxaparin 40 mg per day (Active Comparator)
  Interventions: Drug: Enoxaparin
- Enoxaparin 1 mg per kg daily (Active Comparator)
  Interventions: Drug: Enoxaparin
- Pre prescribed regimen of Enoxaparin (Active Comparator): Current enoxaparin dose at time of first prenatal visit.
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Drug: Enoxaparin 40 mg every morning until 36 weeks gestation. Drug: Enoxaparin 1 mg per kg every morning until 36 weeks gestation. Dose will increase at wt. increases.
  Drug: Enoxaparin dose taken by patient when enrolled until 36 weeks gestation.

SUMMARY:
Enoxaparin is a type of low molecular weight heparin (LMWH), or anticoagulant, used to prevent and treat blood clots. Formation of blood clots, or venous thromboemboli (VTE) in pregnancy can have dangerous and even life-threatening effects on the mother and fetus. Enoxaparin is the preferred medicine to prevent clotting in pregnant patients who are at risk for VTE, because it has been studied to be safe and effective in pregnancy without any harms to the fetus. Although this medication is routinely used and is recommended by several prominent medical groups, the optimal dosing for prevention of VTE is still unclear. The range of standardly prescribed dosing regimens of Enoxaparin includes 40mg daily and 1mg/kg daily, but these two dosing strategies have never been compared in a head to head fashion.

DETAILED DESCRIPTION:
When pregnant patients are diagnosed by their physician as being at risk for VTE, or when they enter the perinatology practice on a previously-prescribed prophylactic enoxaparin regimen, they will be offered a chance to discuss participation in the study. The patient will be consented and those who are not already receiving enoxaparin will be prescribed one of the two dosing regimens, at their physician's discretion, at that same clinic visit.

A baseline blood sample will be drawn to assess coagulation using thromboelastography [TEG]. TEG is a point-of-care device which measures the viscoelastic properties of clot formation. This device can provide rapid and detailed information about coagulation changes. TEG will be used to assess coagulation changes after commencing treatment with enoxaparin (see later).

As per routine care, the patient will be instructed by the clinic nurse on how to fill her prescription at the pharmacy, how to give herself the injection subcutaneously once daily in the morning, and how to troubleshoot the injection process. As per routine care, the patient will have the opportunity to ask all questions necessary about this process, and her understanding and ability to comply with the injection procedures will be assessed by the clinic RN. The patient will be given a new prescription as needed by her physician at her regularly scheduled MD appointment. At any time, as per routine care, the patient can have the opportunity to review or troubleshoot the injection process with the RN or MD in the clinic. At each clinic visit, as per routine care, approximately 1-2 times per month as per routine care, the patient will be weighed and her weight recorded in her prenatal chart. At each of these visits the patient will also be asked a series of questions as per the study flowsheet in the chart, about potential side effects or adverse events she may have experienced since her last visit. In addition, she will receive a phone call from one of the study investigators once to twice per month to enquire about side effects, medication tolerability, and medication compliance. At 3 predetermined intervals throughout the pregnancy, the patient will be instructed to give a blood sample at the outpatient laboratory. When at all possible, these blood draws will be coordinated to coincide with the patient's regularly scheduled prenatal care blood draws, to minimize venipuncture episodes. The study blood sample results will test for: anti-Xa level , which is a marker of the effective prophylactic range of Enoxaparin, serum creatinine, which is a marker of kidney function and renal clearance of medication, and also for coagulation analysis (using TEG) to assess the coagulation effects of enoxaparin. TEG is a point-of-care device which measures the viscoelastic properties of clot formation. This device can provide rapid and detailed information about coagulation changes. The anti-XA level sample results will be blinded to the medical care providers and to the patient, and used for research purposes only. At or shortly after the patient reaches 36 weeks gestation, she will be switched from enoxaparin to unfractionated heparin (UFH), as per standard of care to avoid any potentially unexpected bleeding events associated with the onset of labor at term. When the patient comes to the hospital for Labor and Delivery, routine labor and delivery care will ensue at the discretion of the medical care team. 24 hours after delivery, or at the discretion of the medical care team, the patient will be restarted on her Enoxaparin dosing arm, as per standard of care. She will be instructed to continue the enoxaparin for 6 weeks, and will receive a prescription from the in-hospital providers for this. The patient will return for a 6 week follow-up visit in the clinic as per standard of care, and a final study blood draw will be performed at that time.

If the patient misses her 6 week appointment, she will receive a phone call to reschedule as per standard of care, and will be instructed over the phone to discontinue her Enoxaparin and to come in for a blood draw.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Warrants prophylaxis against venous thromboembolism in pregnancy according to American College of

Obstetrics and Gynecology Practice Bulletin 2000, reaffirmed in 2008:

* history of idiopathic thrombosis
* history of thrombosis related to pregnancy or oral contraceptive use
* history of thrombosis accompanied by an underlying thrombophilia other than homozygous for the factor V Leiden mutation, heterozygous for both the factor V Leiden and the prothrombin G20210A mutation, or AT-III deficiency
* without a history of thrombosis but who have an underlying thrombophilia and a strong family history of thrombosis
* Known thrombophilia except for those listed above, with a history of adverse pregnancy outcome (APO) as defined by: ¡Ý3 pregnancy losses in the 1st trimester, ¡Ý2 pregnancy losses/stillbirth in 2nd trimester, ¡Ý1 pregnancy loss/intrauterine fetal demise (IUFD) in the 3rd trimester, intrauterine growth restriction (IUGR), abruptio placentae, or severe pre-Eclampsia prior to 34 weeks gestation.

Exclusion Criteria:

1. Need for therapeutic-level anticoagulation as determined by physician
2. Renal disease as defined by serum creatinine >1.0
3. Weight >90kg
4. Allergy to enoxaparin

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-05; Primary Completion 2011-08 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Judith Lyell, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Middleton P, Shepherd E, Gomersall JC. Venous thromboembolism prophylaxis for women at risk during pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2021 Mar 29;3(3):CD001689. doi: 10.1002/14651858.CD001689.pub4. PMID 33779986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 11/2/09 to 1/13/11 in the Obstetric Clinic at Lucile Packard Children's Hospital.
Pre-assignment Details: There were no significant events.
Groups:
- Enoxaparin 40 mg Per Day: 40 mg Enoxaparin injection daily
- Enoxaparin 1 mg Per kg Daily: 1 mg/kg Enoxaparin injection daily
- Enoxaparin 60 mg Per Day: 60 mg Enoxaparin injection daily - Pre prescribed regimen
Period: Overall Study
Arm/Group | Enoxaparin 40 mg Per Day | Enoxaparin 1 mg Per kg Daily | Enoxaparin 60 mg Per Day
Started | 3 | 6 | 2
Completed | 3 | 6 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants in study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Enoxaparin 40 mg Per Day | Enoxaparin 1 mg Per kg Daily | Enoxaparin 60 mg Per Day | Total
Number analyzed (Participants) | 3 | 6 | 2 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 2 | 11
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (2.1) | 32.8 (6.2) | 34.5 (6.4) | 34.2 (1.04)
Gender [Count of Participants; unit: Participants]
  Female | 3 | 6 | 2 | 11
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 5 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 2 | 0 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 2 | 11
Gestational Age at Enrollment [Mean (Full Range); unit: weeks] | 10.86 [7.71 to 12.71] | 12.19 [10.00 to 15.29] | 11.64 [9.86 to 13.43] | 11.73 [7.71 to 15.29]
Weight at Enrollment [Mean (Full Range); unit: kg] | 61.7 [57 to 69] | 65.5 [54 to 83] | 59.5 [59 to 60] | 63.4 [54 to 83]
BMI at Enrollment [Mean (Full Range); unit: kg/m2] | 22.8 [20.9 to 23.7] | 26.3 [18.4 to 34.6] | 22.6 [21.4 to 23.9] | 24.7 [18.4 to 34.6]
Insurance Status [Number; unit: participants]
  Public | 0 | 2 | 0 | 2
  Private | 3 | 4 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Peak Anti-Xa Level
Description: Goal peak anti-Xa level is 0.2 to 0.4 u/ml. We compared peak drug levels between different dosing arms.
Time Frame: One measurement per trimester of pregnancy, up to 36 weeks
Measure: Mean (Standard Deviation); unit: u/ml
Arm/Group | Enoxaparin 40 mg Per Day | Enoxaparin 1 mg Per kg Daily | Enoxaparin 60 mg Per Day
Number analyzed (Participants) | 3 | 6 | 2
u/ml
  14-18 weeks gestation | 0.35 (0.07) | 0.46 (0.27) | 0.57 (0.01)
  24-28 weeks gestation | 0.27 (0.1) | 0.34 (0.23) | 0.34 (0.1)
  32-34 weeks gestation | 0.22 (0) | 0.55 (0.23) | 0.56 (0.07)
Statistical Analysis 1: Comparison: Enoxaparin 40 mg Per Day vs Enoxaparin 1 mg Per kg Daily vs Enoxaparin 60 mg Per Day; at 14-18 weeks gestational age; Test type: Superiority or Other; p = 0.4, Kruskal-Wallis
Statistical Analysis 2: Comparison: Enoxaparin 40 mg Per Day vs Enoxaparin 1 mg Per kg Daily vs Enoxaparin 60 mg Per Day; at 24-28 weeks gestational age; Test type: Superiority or Other; p = 0.9, Kruskal-Wallis
Statistical Analysis 3: Comparison: Enoxaparin 40 mg Per Day vs Enoxaparin 1 mg Per kg Daily vs Enoxaparin 60 mg Per Day; at 32-34 weeks gestational age; Test type: Superiority or Other; p = 0.3, Kruskal-Wallis

2. Secondary Outcome: Thromboembolic Events
Time Frame: Enrollment through 6 weeks postpartum
Measure: Number; unit: participants
Arm/Group | Enoxaparin 40 mg Per Day | Enoxaparin 1 mg Per kg Daily | Enoxaparin 60 mg Per Day
Number analyzed (Participants) | 3 | 6 | 2
participants | 0 | 0 | 0

3. Secondary Outcome: Bleeding Events
Time Frame: Enrollment through 6 weeks postpartum
Measure: Number; unit: participants
Arm/Group | Enoxaparin 40 mg Per Day | Enoxaparin 1 mg Per kg Daily | Enoxaparin 60 mg Per Day
Number analyzed (Participants) | 3 | 6 | 2
participants | 1 | 0 | 0

4. Secondary Outcome: Side Effect - Bruising
Time Frame: Enrollment through 6 weeks postpartum
Measure: Number; unit: participants
Arm/Group | Enoxaparin 40 mg Per Day | Enoxaparin 1 mg Per kg Daily | Enoxaparin 60 mg Per Day
Number analyzed (Participants) | 3 | 6 | 2
participants | 1 | 3 | 0

ADVERSE EVENTS:
Time Frame: Enrollment through 6 weeks postpartum.
Arm/Group | Enoxaparin 40 mg Per Day | Enoxaparin 1 mg Per kg Daily | Enoxaparin 60 mg Per Day
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 0/2

LIMITATIONS AND CAVEATS:
Small numbers of subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No